CLINICAL TRIAL: NCT04945356
Title: The Use of Telerehabilitation to Improve Function and Quality of Life for People in the Chronic Phase After Stroke During Pandemic Containment Measures of COVID19 : a Feasibility Pilot Study
Brief Title: Telerehabilitation During Pandemic Containment Measures of COVID19
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: McGill University (Other); Université du Québec à Chicoutimi (Other); Université de Montréal (Other)
Responsible Party: Principal Investigator, Marie-Hélène Milot, researcher and principal investigator, Université de Sherbrooke
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MP-31-2021-3817
Record Dates: First submitted 2021-06-24; First posted 2021-06-30 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Stroke
Keywords: stroke; telerehabilitation; COVID19; function; upper limb; quality of life
MeSH Terms: conditions — Stroke; COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- upper limb virtual training (Experimental): 6-week virtual training of the affected upper limb using the Physiotec application
  Interventions: Other: upper limb training

INTERVENTIONS:
Other: upper limb training — The 6-week exercise program will consist of evidence-based exercises covering the breadth and depth of rehabilitation interventions. The therapist will choose the appropriate exercises for each participant's level of function from more than 15,000 exercises implemented within the Physiotec app and developed by rehabilitation experts. Personalized upper limb exercises will be based on the therapist initial assessment of participants, using the TERA+ telerehabilitation platform, and their goals. After each training session, participants will have to rate their perceived level of effort on a Borg scale (/10). The Borg scores will be monitored by the therapist as a precautionary measure to ensure safety and appropriateness of intensity of exercises. Participants will be instructed to train at a target score of around 7/10 (somewhat hard) on the Borg scale.

SUMMARY:
BACKGROUND:

Although rehabilitation is effective in restoring function, many elderly individuals, especially those who have survived a stroke, are no longer receiving adequate rehabilitation services during the COVID19 pandemic due to containment measures. To overcome this problem, telerehabilitation is a promising avenue to deliver customized and personalized at-home therapy sessions while adhering to physical distancing guidelines.

OBJECTIVES:

The primary objective of this study is to evaluate the feasibility of using customized and personalized at-home therapy sessions using the Physiotec application for individuals with a stroke. A second objective is to measure the potential efficacy of the telerehabilitation intervention at improving function and quality of life based on standardized clinical measures and measures of improvement implemented in the Physiotec application.

METHODS:

We propose a non-randomized, single-group trial. Twenty-five individuals will be recruited on a voluntary basis. To be included, participants must 1) be ≥18 years old; 2) have a single unilateral stroke (≥ 6 months); 3) have minimal return of function in the affected upper limb; and 4) no longer be receiving rehabilitation treatments. Participants will receive a tablet containing the Physiotec application training program and TERA+, a telerehabilitation platform. The training program of the affected upper limb will last 6 weeks (90 minutes/week) and will be updated 3 times (weeks 1-3-5) by the therapist, using the TERA+ platform, based on the participant's functional capacity and progress, as measured by the app. Feasibility will be assessed by means of retention rate, adverse events, adherence to the telerehabilitation intervention, satisfaction with its use and with the exercise program. Efficacy will be assessed by several questionnaires on life habits, motor recovery and quality of life.

RELEVANCE:

This study will inform as to the optimal delivery of adapted rehabilitation services for stroke survivors that are currently not receiving optimal rehabilitation services because of the ongoing COVID19 pandemic. The results will serve to support in-home rehabilitation exercises aimed at promoting recovery, independent living and improving quality of life for stroke survivors.

ELIGIBILITY:
Inclusion Criteria:

1. be over 18 years of age;
2. present a single unilateral stroke for more than 6 months;
3. have a minimal motor return to the upper limb assessed visually via the visuo-conference platform;
4. no longer receiving any in- or outpatient rehabilitation services.

Exclusion Criteria:

1. severe spasticity that prevents movement of the affected limb (score > 3 on the modified Ashworth scale);
2. an orthopedic problem with the affected upper limb or lower limb;
3. any neurological problem other than that arising from a stroke;
4. cognitive impairment (a score ≤ 2/5 on the Mini-Cog Test);
5. fall that has required physician evaluation within the past six months;
6. other neurologic, neuromuscular, or orthopedic disease or comorbidities that would prevent exercise participation or increase participant risk;
7. vision or hearing, communication, literacy or perceptual impairment that would interfere with app use as assessed by the study physical therapist during the screening process through a direct demonstration of the app and try out of the app

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2020-10-28 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Retention rate to the telerehabilitation intervention | in the week after the last session of telerehabilitation training
  the number of participants enrolled at the end of the study divided by the number of participants recruited at the beginning of the study
Adherence to the telerehabilitation training program | in the week after the last session of telerehabilitation training
  the number of telerehabilitation training sessions that participants took part in during the 6-week training program
Adverse events related to the intensity of training assessed with the Borg scale embedded within the Physiotec application | after each training session throughout the duration of the telerehabilitation training program
  Adverse events related to the intensity of training will be tracked after each training session via the BORG scale (intensity of training should not be done at a score higher than 7/10)
Adverse events related to pain levels assessed with the visual analog scale embedded within the Physiotec application | after each training session throughout the duration of the telerehabilitation training program
  Adverse events related to pain will be tracked after each training session with a 0-10 visual analog scale for pain (training will be adjusted if pain score is greater than 7/10).
Participants' satisfaction with telerehabilitation assessed with the Telerehabilitation Satisfaction questionnaire | in the week after the last session of telerehabilitation training
  Telerehabilitation Satisfaction questionnaire: this questionnaire contains 15 questions where the participants rate their satisfaction about the use of telerehabilitation on a Likert scale (from strongly agree to strongly disagree or undecided).
Participants' satisfaction with the application assessed with the User Satisfaction questionnaire | in the week after the last session of telerehabilitation training
  User Satisfaction questionnaire: this questionnaire contains 6 questions about the participants satisfaction about the application (from 1 = not at all to 5 = extremely)
Participants' satisfaction with the exercise program assessed with the Health Care Satisfaction questionnaire | in the week after the last session of telerehabilitation training
  Health Care Satisfaction questionnaire: this questionnaire comprises 26 questions about the participants feeling (from 1= not at all to 4= extremely) and the importance they give to different situations (from 1= not important to 4 = extremely important) related to the training program

SECONDARY OUTCOMES:
Change in quality of life assessed with the 12-item Short Form Survey | baseline and in the week after the last session of telerehabilitation training
  SF-12: this 12-question health survey assesses both physical and mental components of the respondent's current health status compared to their health status one month ago. It covers 8 domains such as limitations in physical activities because of health problems and bodily pain. Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning.
Change in life habits assessed with the LIFE-H 3.0 questionnaire | baseline and in the week after the last session of telerehabilitation training
  LIFE-H 3.0: this test includes 240 items and assesses the level of participation in daily activities and social roles. It also considers the degree of difficulty in carrying out tasks as well as the type of assistance required by the person. Each question is scored on a 0-9 scale where a score of 0 implies a total disruption of participation.
Change in the quantity and quality of affected upper limb use assessed with the Motor Activity Log | baseline and in the week after the last session of telerehabilitation training
  Motor Activity Log-14: this questionnaire assesses, on a 6-point ordinal scale, the use and quality of use of the affected upper limb in 14 everyday activities. A high score means that the participant perceives a greater use of his arm and a better quality of movement.
Change in reintegration to social activities assessed with the Reintegration to Normal Living Index | baseline and in the week after the last session of telerehabilitation training
  Reintegration to Normal Living Index: this questionnaire covers the following domains: indoor, community, distance mobility, self-care, daily activity, recreational and social activities, family role(s), personal relationships, presentation of self to others and general coping skills. Using 11 questions, it quantitatively assesses, on a 0-10 cm visual analogue scale, the degree to which individuals achieve reintegration into normal living. Each score is summed to provide a total score out of 110 points (adjusted back to 100) where a higher score indicates a better perception of reintegration
Change in motor recovery of affected upper limb assessed with the Stroke Rehabilitation Assessment of Movement | baseline and in the week after the last session of telerehabilitation training
  Stroke Rehabilitation Assessment of Movement: it is a performance-based measure that evaluates, on a 3-point ordinal scale, motor recovery at the affected upper limb. The total score for the upper limb section is 20 points with a higher score indicating a better motor recovery.
Change in range of motion at the affected upper limb assessed visually | baseline and in the week after the last session of telerehabilitation training
  Range of motion of the upper extremity will be visually estimated by a research assistant, using the TERA+ platform, for the shoulder (flexion), elbow (flexion & extension), forearm pronation/supination, wrist (extension & flexion) and finger (flexion & extension).
Participants' perceived improvement of the affected upper limb following training assessed with the Global Rating of Change Score questionnaire | in the week after the last session of telerehabilitation training
  Global Rating of Change Score: this questionnaire will assess the participant's perceived improvement in the function of his trained upper limb on a 7-point ordinal scale from 3 (very much improved) to -3 (very much worse)
Fear of COVID assessed with the Fear of COVID-19 scale | baseline
  Fear of COVID-19 scale: this 7-item questionnaire will assess the perception of the participants about the COVID19 pandemic using a five-item Likert- type scale (from "strongly disagree" to "strongly agree"). The minimum score possible for each question is 1, and the maximum is 5. A total score is calculated by adding up each item score. The higher the score, the greater the fear of coronavirus-19 is.

CONTACTS AND LOCATIONS:
Locations (3):
- Canada (3):
  - Université du Québec à Chicoutimi, Chicoutimi, Quebec
  - McGill University, Montreal, Quebec
  - Centre de recherche sur le vieillissement, Sherbrooke, Quebec

IPD SHARING:
Plan to Share IPD: No